CLINICAL TRIAL: NCT00701194
Title: Early Intervention Foster Care: A Prevention Trial
Acronym: EIFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Philip A. Fisher, PhD, Study Principal Investigator, Oregon Social Learning Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH059780 (NIH)
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: School Readiness; Developmental Delays
Keywords: placement instability; disruptive behavior disorders; school readiness; developmental delays; cortisol; executive functioning; therapeutic foster care; prevention; early intervention
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): EIFC/MTFC-P
  Interventions: Behavioral: Early Intervention Foster Care (EIFC)
- 2 (No Intervention): Services as usual
- Community Comparison (No Intervention): Non-maltreated community pre-schoolers from low-income biological families.

INTERVENTIONS:
Behavioral: Early Intervention Foster Care (EIFC) — The EIFC/MTFC-P intervention is delivered through a treatment team approach. Foster parents receive preservice training and ongoing consultation from program staff. Children receive individual therapy and attend a therapeutic playgroup. The intervention emphasizes the use of concrete encouragement for prosocial behavior; consistent, nonabusive limit-setting to address disruptive behavior; and close supervision of the child. The EIFC intervention employs a developmental framework in which the challenges of foster preschoolers are viewed from the perspective of delayed maturation and is oriented toward creating optimal environmental conditions to facilitate developmental progress. These conditions include a responsive and consistent caregiver and a predictable daily routine.
  Other Names: Multidemensional Treatment Foster Care-Preschool (MTFC-P)
  Arms: 1

SUMMARY:
The Early Intervention Foster Care [EIFC] project is an efficacy trial of the Oregon Social Learning Center Multidimensional Treatment Foster Care Program, a preventive intervention that targets 3 commonly co-occurring variables among young foster children: (1) behavioral problems, (2) physiological dysregulation within the neuroendocrine system (i.e., HPA axis activity), and (3) developmental delays.

DETAILED DESCRIPTION:
The Early Intervention Foster Care project is an ongoing randomized efficacy trial to evaluate the Early Intervention Foster Care Program (EIFC). EIFC, also known at Multidimensional Treatment Foster Care-Preschool (MTFC-P), is a preventive intervention that is specifically designed to address the needs of preschool-aged foster children and their caregivers. Over the first 5 years of the project data was collected from 177 preschool-aged children, 117 of whom were in the Oregon foster care system and 60 of whom were living with their biological families for a community comparison sample. Foster children in the study were randomly assigned to the EIFC experimental intervention condition or a regular foster care condition (RFC). The following hypotheses are under investigation: (1) Relative to children in the RFC condition, children in the EIFC condition will show greater improvements in temporally proximal outcomes (e.g., behavioral/emotional, salivary cortisol, and developmental) and in temporally distal outcomes (e.g., behavioral functioning in the school setting; long-term placement stability, including reunification or adoption; and mental health status, including psychiatric diagnoses). (2) Proximal outcomes over the course of the intervention will predict distal outcomes during the early elementary school years. (3) Proximal outcomes will be mediated by caregivers' childrearing practices-specifically, engagement with and monitoring of the child in the home, the quality and consistency of parental discipline, and the use of positive reinforcement strategies. (4) The same childrearing practices will mediate the psychosocial adjustment of the child in the aftercare setting (i.e., return to family of origin, placement in adoptive home, or continued placement in long-term foster home). (5) The EIFC intervention will cost-effectively reduce the need for mental health and social services for children, decreasing the length of time that children spend in foster care and reducing the need for special education services for children.

ELIGIBILITY:
Inclusion Criteria:

* child age 3 to 6 years currently in foster care
* child has entered new foster placement
* child currently living in Lane County, Oregon

Exclusion Criteria:

* child is medically or developmentally unable to complete assessment tasks

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 1999-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
placement stability | 6 months to 48 months post-intervention

SECONDARY OUTCOMES:
attachment and behavioral regulation | baseline through 48 months post-intervention
neuroendocrine and executive functioning | baseline through 48 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Fisher, PhD, Principal Investigator — Oregon Social Learning Center
Locations (1):
- Oregon Social Learning Center, Eugene, Oregon, United States

REFERENCES:
- See also: Oregon Social Learning Center website — http://www.oslc.org